CLINICAL TRIAL: NCT06255444
Title: Body Mass Index Patients With Cervical Radiculopathy
Brief Title: Cervical Radiculopathy and Body Mass Index
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Study director, PT, MsC, Karabuk University
Other Study IDs: Karabuk University-06
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Radiculopathy, Cervical
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight/Obese BMI: This group consists of overweight and obese patients diagnosed with cervical radiculopathy by a neurosurgeon.
- Normal BMI: This group consists of patients with normal BMI who were diagnosed with cervical radiculopathy by a neurosurgeon.

SUMMARY:
Body Mass Index (BMI) is thought to impact radiculopathy symptoms. The pressure exerted by fatty tissue on muscle tissue can also significantly affect the nerves. This condition causes radiculopathy. Therefore, high BMI causes an increase in the incidence of radiculopathy. Consequently, it is thought that pain caused by cervical radiculopathy may be related to BMI and affect functionality. Also, it is believed that with the increase in the load on the cervical region, there will be an increase in degenerative disorders and an increase in the incidence of radiculopathy. This study examines the relationship between BMI and peripheral muscle strength, pain, range of motion, disability, quality of life, and functionality in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
When radiculopathy occurs due to compression of the neck nerve roots due to pathologies in the neck, it is called cervical radiculopathy. It is thought that high and low BMI values have an impact on radiculopathy. The pressure exerted by fatty tissue on muscle tissue can significantly affect the nerves. This causes an increase in radiculopathy symptoms. Therefore, high BMI causes an increase in the incidence of radiculopathy. The relationship between the degree of obesity, visceral fat area, body mass index, abdominal circumference, and lumbar disc herniation and pain is shown. It has been stated in the literature that BMI is related to lumbar radiculopathy and pain level. Still, there appear to be inadequacies in examining its relationship with radiculopathy, which is related to upper extremity functionality. Therefore, it is thought that pain caused by cervical radiculopathy may be associated with BMI and affect functionality more. At the same time, as BMI increases, lumbar lordosis may affect spine biomechanics, leading to deterioration in sagittal balance and an increase in cervical problems. According to an international study It is stated that in obese individuals with high BMI values, vertebral discs undergo degeneration due to the load on the spine.

For this reason, researchers have suggested that pain level increases linearly with BMI value. It is stated that degenerating lumbar vertebrae progress to narrowing over time and that the risk of lumbar spinal stenosis may increase in individuals with high-fat content. Therefore, radiculopathy is thought to be a significant factor when looking at the relationship between pain in the musculoskeletal system and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having cervical pathology detected by a neurosurgeon with MRI and having radicular pain symptoms related to this
* BMI >18.5 kg/m2
* Having symptoms for at least 3 months
* Being able to communicate in Turkish
* Volunteering to participate in the study.

Exclusion Criteria:

* Pregnant patients
* Presence of malignancy in the spine
* Having a serious neurological disease
* Primary or metastatic spinal malignancy, history of spinal fractures
* People with neurological diseases (Hemiplegia, Multiple Sclerosis, Parkinson, etc.).
* Being diagnosed with advanced osteoporosis
* Having undergone a surgical intervention involving the cervical region within the last year
* Lack of cooperation

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Normal, overweight and obese patients with cervical radiculopathy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity | First Day
  A visual analog scale will be used to evaluate individuals' neck and arm pain levels during rest and activity.
Disability | First Day
  "Neck Disability Index" (NDI) will be used to evaluate the effects of neck pain on daily living activities. The scale is scored between 0 and 100, and a higher score indicates higher disability.
Range of Motion | First Day
  A universal goniometer will be used to evaluate the flexion and extension cervical region joint range of motion of the patients.
Peripheral Muscle Strength | First Day
  Shoulder abduction and shoulder flexion muscle strength will be measured by using hand-held dynamometer.
Grip strength | First Day
  Hand grip strength will be measured by using Jamar Hand Dynamometer
Qulity of life | The scale is scored between 0-100, and a higher score indicates an increase in quality of life.
  Short Form-36 will be used to determine the quality of life level.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Güneş, MsC, Study Director — Deparment of Physical Therapy and Rehabilitation, Faculty of Health Sciences, Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mateos-Valenzuela AG, Gonzalez-Macias ME, Ahumada-Valdez S, Villa-Angulo C, Villa-Angulo R. Risk factors and association of body composition components for lumbar disc herniation in Northwest, Mexico. Sci Rep. 2020 Oct 28;10(1):18479. doi: 10.1038/s41598-020-75540-5. PMID 33116248
- [Result] Stienen MN, Joswig H, Smoll NR, Corniola MV, Schaller K, Hildebrandt G, Gautschi OP. Influence of Body Mass Index on Subjective and Objective Measures of Pain, Functional Impairment, and Health-Related Quality of Life in Lumbar Degenerative Disc Disease. World Neurosurg. 2016 Dec;96:570-577.e1. doi: 10.1016/j.wneu.2016.09.070. Epub 2016 Sep 28. PMID 27686509
- [Result] Sheng B, Feng C, Zhang D, Spitler H, Shi L. Associations between Obesity and Spinal Diseases: A Medical Expenditure Panel Study Analysis. Int J Environ Res Public Health. 2017 Feb 13;14(2):183. doi: 10.3390/ijerph14020183. PMID 28208824